CLINICAL TRIAL: NCT04399460
Title: The Effects of Long-term Consumption of Full-fat Dairy Products on Satiety, Body Weight and Glycemic Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFC_LTDairy_2019
Record Dates: First submitted 2020-05-12; First posted 2020-05-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Overweight or Obesity; Body Weight
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dairy Energy Restrictive Diet (Experimental): Low-dairy (<1 serving/day) and 500kcal/deficit per day energy restrictive diet
  Interventions: Other: Restrictive Eating
- 3 Servings of Full-Fat Dairy with Energy Restrictive diet (Experimental): Energy-restrictive diet (500 kcal/deficit per day) with 3 servings of full-fat dairy products from full-fat milk, and assorted yogurts and cheeses
  Interventions: Other: Dairy-based commercially available food products; Other: Restrictive Eating
- 3 Servings of Full-Fat Dairy but no energy restriction (Experimental): Normal diet (no energy restriction) with 3 servings of full-fat dairy products from full-fat milk, and assorted yogurts and cheeses
  Interventions: Other: Dairy-based commercially available food products

INTERVENTIONS:
Other: Dairy-based commercially available food products — Full-fat milk (3.25% milk, 250 mL), assortment of yogurts, and cheeses
  Arms: 3 Servings of Full-Fat Dairy but no energy restriction; 3 Servings of Full-Fat Dairy with Energy Restrictive diet
Other: Restrictive Eating — Dietitian will assist with 500 kcal/day reduction through limiting of macronutrients 45-65% energy from carbohydrates 20-35% energy from fat 10-35% energy from protein
  Arms: 3 Servings of Full-Fat Dairy with Energy Restrictive diet; Low Dairy Energy Restrictive Diet

SUMMARY:
The proposed study looks at the effect of long-term diet modification with or without full-fat dairy products or restrictive eating on body weight, body composition and cardiometabolic markers in healthy overweight/obese men and women.

DETAILED DESCRIPTION:
A total of 93 males and females will participate in the study at the University of Toronto.

At the beginning and after 12 weeks, body weight, composition will be measured through Bodpod scans. Resting metabolic rate and thermogenesis will be measured by indirect calorimetry. Also, fecal samples will be collected for gut microbiome profiling along with blood for glucose, insulin, hormones, triacylglycerol, HbA1c, short-chain fatty acid, red blood cells and FGF21. Urine samples will be collected throughout the study.

A followup session at 16 weeks will reassess previous measures.

ELIGIBILITY:
Inclusion Criteria:

* BMI: ≥ 27 and ≤ 34.9 kg/m2
* Fasting serum glucose: ≤ 7 mmol/L
* Low ≤1 serving of dairy consumption
* Waist circumference >88cm (women) and >102cm (men)
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Willing to maintain current dietary supplement use throughout the trial. On test days, participant agrees not to take any dietary supplements until dismissal from the study. Failure to comply will result in a rescheduled test visit.
* Willing to abstain from alcohol consumption for 24 h prior to all test visits.
* Willing to avoid vigorous physical activity for 24 h prior to all test visits.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator

Exclusion Criteria:

* Fasting blood glucose > 7 mmol/L
* Triglycerides ≥ 2.3 mmol/L
* Smoking tobacco products and marijuana
* Thyroid problems
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, any malabsorptive syndrome, pancreatitis, gallbladder or biliary disease.
* Presence of gastrointestinal disorder or surgeries within the past year.
* Consuming prescription or non-prescription drug, herbal or nutritional supplements known to affect blood glucose or that could affect the outcome of the study as per investigator's judgement.
* Known to be pregnant or lactating, or planning on becoming pregnant in the next 12 months.
* Irregular menstrual cycles (i.e. frequent missed cycles), menopausal or post- menopausal
* Unwillingness or inability to comply with the experimental procedures
* Known intolerance, sensitivity or allergy to dairy products
* Consumption of protein powders/protein supplements
* Extreme dietary habits
* Uncontrolled hypertension as defined by the average blood pressure measured at screening.
* Weight gain or loss of at least 10 lbs in previous three months, and history of childhood overweight or obesity
* Excessive alcohol intake
* Restrained Eaters

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Starting at the beginning of the study 0 week then biweekly for 7 sessions up to 12 weeks with a followed up at 16 weeks.
  Each participant will attend 8 sessions biweekly in total

OTHER OUTCOMES:
Fecal Collection | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Gut microbiome profiling
Change in blood glucose levels | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total
Change in fasting insulin (µIU/mL) levels in the blood | Change from baseline at 12 weeks
  Each participant will attend 3 sessions in total
Change in gut hormone levels measured in the blood | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total
Change in triacylglycerol level (mg/dL) | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total
Change in HbA1c (mmol/mol) | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total
Change in red blood cells fatty acids | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total
Change in resting metabolic rate | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total measured by Indirect calorimetry
Change in short-chain fatty acids in the blood | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total
Change in waist and hip circumference in cm | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total
Change in lean body mass percentage measured by BodPod | Starting at the beginning of the study 0 week then at 12 weeks with a followed up at 16 weeks.
  Each participant will attend 3 sessions in total

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Mount Saint Vincent University, Halifax, Nova Scotia
  - Department of Nutritional Sciences, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderson GH, Chen Zhou CZ, Vien S, Soo M, Salamat S, Akbarifakhrabadi M, Chomka L, Kathirvel P, Siddiqi F, Fabek H, Luhovyy B. The effect of three daily servings of full-fat dairy for 12 weeks on body weight, body composition, energy metabolism, blood lipids, and dietary intake of adults with overweight and obesity. J Nutr. 2026 Jan 22:101373. doi: 10.1016/j.tjnut.2026.101373. Online ahead of print. PMID 41580085